CLINICAL TRIAL: NCT06606808
Title: Investigating the Safety, Feasibility, and Optimal Dose of Risankizumab-800CW for Visualizing Drug Targeting in Inflammatory Bowel Disease
Brief Title: Fluorescence Imaging of Risankizumab-800CW in Inflammatory Bowel Disease
Acronym: NAVIGATE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: UMCG 20010; 2024-515358-25-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-10; First posted 2024-09-23 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis (UC); Crohn Disease (CD)
Keywords: Fluorescence Molecular Endoscopy; Inflammatory Bowel Disease; Risankizumab-800CW
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 4.5 mg risankizumab-800CW (Experimental): Patients receive 4.5 mg risankizumab-800CW and undergo a Fluorescence Molecular Imaging procedure
  Interventions: Drug: Risankizumab-800CW 4.5 mg
- 15 mg risankizumab-800CW (Experimental): Patients receive 15 mg risankizumab-800CW and undergo a Fluorescence Molecular Imaging procedure
  Interventions: Drug: Risankizumab-800CW 15 mg
- 25 mg risankizumab-800CW (Experimental): Patients receive 25 mg risankizumab-800CW and undergo a Fluorescence Molecular Imaging procedure
  Interventions: Drug: Risankizumab-800CW 25 mg
- 14 weeks or more of risankizumab therapy and optimal dose risankizumab-800CW (Experimental): Patients who are treated with risankizumab for at least 14 weeks are enrolled in this arm. This can be patients who already joined in the dose finding part of the study or new patients. These patients will receive the optimal dose risankizumab-800CW and will undergo aFluorescence Molecular Imaging procedure
  Interventions: Drug: Risankizumab-800CW optimal dose

INTERVENTIONS:
Drug: Risankizumab-800CW 4.5 mg — Risankizumab-800CW will be administered intravenously. 2-3 days later, a Fluorescence Molecular Imaging procedure will be performed to enable the visualisation and detection of fluorescence signals.
  Arms: 4.5 mg risankizumab-800CW
Drug: Risankizumab-800CW 15 mg — Risankizumab-800CW will be administered intravenously. 2-3 days later, a Fluorescence Molecular Imaging procedure will be performed to enable the visualisation and detection of fluorescence signals.
  Arms: 15 mg risankizumab-800CW
Drug: Risankizumab-800CW 25 mg — Risankizumab-800CW will be administered intravenously. 2-3 days later, a Fluorescence Molecular Imaging procedure will be performed to enable the visualisation and detection of fluorescence signals.
  Arms: 25 mg risankizumab-800CW
Drug: Risankizumab-800CW optimal dose — Risankizumab-800CW will be administered intravenously. 2-3 days later, a Fluorescence Molecular Imaging procedure will be performed to enable the visualisation and detection of fluorescence signals.
  Arms: 14 weeks or more of risankizumab therapy and optimal dose risankizumab-800CW

SUMMARY:
Crohn's Disease (CD) and Ulcerative Colitis (UC) are chronic inflammatory bowel diseases (IBD). Risankizumab is a human monoclonal antibody against IL23 p19, part of a pro-inflammatory cytokine that mediates the inflammatory response in IBD upon binding to its receptor. Primary non-response to risankizumab is high in both CD and UC. Currently, there are no predictors of response to risankizumab and the actual mechanism of action has not yet been elucidated. To gain better understanding of the drug targeting of risankizumab in IBD, the University Medical Center Groningen (UMCG) developed fluorescently labeled risankizumab (risankizumab-800CW). This study aims to assess the safety and the optimal dose of risankizumab-800CW to visualize and potentially quantify the local drug concentration and predict treatment response in IBD patients using in vivo and ex vivo fluorescence molecular imaging (FMI).

ELIGIBILITY:
Inclusion Criteria for part A:

* Established IBD diagnosis
* Active disease: clinically active disease of the bowel is defined clinically as at least mild activity using dedicated scoring indices or biochemically active disease as defined by a fecal calprotectin > 60 μg/g
* Patients must be eligible for risankizumab therapy
* Minimum age of 18 years
* Written informed consent
* Clinical indication for an endoscopic procedure

Inclusion Criteria for part B:

* Established IBD diagnosis
* Patients must be on risankizumab therapy for at least 14 weeks
* Minimum age of 18 years
* Written informed consent
* Clinical indication for an endoscopic procedure

Exclusion Criteria for part A:

* A female study patient who is pregnant or provides breastfeeding
* A female study patient of premenopausal age who does not use any reliable form of contraception at the time of risankizumab-800CW administration and the following 10 weeks
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent
* Prior anti-IL23-specific therapy (IL23/IL12 combination therapy is not an exclusion criteria)
* Active extra gastrointestinal manifestations of Crohn's disease (e.g. uveitis or pyoderma gangrenosum at vital locations)

Exclusion Criteria for part B:

* A female study patient who is pregnant or provides breastfeeding
* A female study patient of premenopausal age who does not use any reliable form of contraception at the time of risankizumab-800CW administration and the following 10 weeks
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent
* Active extra gastrointestinal manifestations of Crohn's disease (e.g. uveitis or pyoderma gangrenosum at vital locations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Determine the safety of risankizumab-800CW in IBD | 2-3 days after administration (day of FME procedure)
  Evaluating possible (severe) adverse events (SAE and AEs)
Blood pressure | Five minutes before, and five and sixty minutes after tracer administration
  Systolic and diastolic in millimeters of mercure (mmHg)
Heart rate | Five minutes before, and five and sixty minutes after tracer administration
  Beats per minute
Temperature | Five minutes before, and five and sixty minutes after tracer administration
  Degrees Celsius
Investigate the feasibility of using ex vivo FMI to detect risankizumab-800CW | 12 months
  Evaluating the performance of ex vivo FMI for detecting risankizumab-800CW signals. This evaluation will be based on mean fluorescence intensities (MFIs) of biopsies and fluorescence/light sheet microscopy.
Investigate the feasibility of using FME to detect risankizumab-800CW signals_1 | 12 months
  Evaluating the performance of FME for detecting risankizumab-800CW signals. This evaluation will be based on MDSFR/SFF measurements.
Investigate the feasibility of using FME to detect risankizumab-800CW signals_2 | 12 months
  Evaluating the performance of FME for detecting risankizumab-800CW signals. This evaluation will be based on a visual evaluation during FME (visible signal yes/no).
Investigate the feasibility of using FME to detect risankizumab-800CW signals_3 | 12 months
  Evaluating the performance of FME for detecting risankizumab-800CW signals. This evaluation will be based on TBR/CNR calculations.
Determining the optimal imaging dose of risankizumab-800CW | 12 months
  The optimal dose will be based on the risankizumab-800CW signals during FME and ex vivo FMI

SECONDARY OUTCOMES:
Investigate a potential correlation of in vivo fluorescence signal intensities and target saturation to clinical response/remission after 14 weeks of risankizumab therapy regimen in patients with IBD | 12 months
  Evaluation of the potential correlation in vivo will be based on in vivo fluorescence images and the MDSFR/SFF measurements before and after at least 14 weeks of risankizumab treatment
Investigate a potential correlation of ex vivo fluorescence signal intensities and target saturation to clinical response/remission after 14 weeks of risankizumab therapy regimen in patients with IBD | 12 months
  Evaluation of the potential correlation ex vivo will be based on MFIs of biopsies, fluorescence microscopy results, and tracer concentrations inside biopsies before and after at least 14 weeks of risankizumab treatment
Quantify the fluorescence signals of the tracer in vivo by using single-fiber reflectance/single-fiber fluorescence (MDSFR/SFF) spectroscopy and correlate these measurements to tracer dose, in vivo fluorescence intensities and inflammation severity | 12 months
  Quantification of MDSFR/SFF measurements in inflamed tissue compared to measurements in non-inflamed tissue. Positive correlation between MDSFR/SFF measurements and dose/inflammation severity?
To correlate ex vivo fluorescence signals to inflammation severity and tracer dose based on histopathological examination inside the obtained biopsies | 12 months
  Histologically ascertained tissue types (qualitative): Normal (non-inflamed) ileal, colon and rectal tissue inflamed ileum, colon and rectum tissue Random ''high-fluorescent'' tissue Random ''Non-fluorescent'' tissue
To assess tracer stability, tracer distribution and tracer concentration, and to identify the composition of immune cells ex vivo to learn more about risankizumab mucosal target cells | 12 months
  Fluorescence (confocal) microscopy with additional use of immune panels and spatial transcriptomics analysis (before and after at least 14 weeks of risankizumab treatment). Measurements of the risankizumab-800CW concentration by light-sheet microscopy after tissue clearing, insights in risankizumab target cells and presence of immune cells inside the biopsies and blood samples by flow cytometry and assessment of tracer stability by Western Blot

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No